CLINICAL TRIAL: NCT05611034
Title: In Vivo Lung Perfusion (IVLP) as an Adjuvant Treatment for Patients With Resectable Pulmonary Metastases of Colorectal Cancers
Brief Title: In Vivo Lung Perfusion (IVLP) for Colorectal Cancer Metastatic to Lung
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-6152
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lung Metastases; Colorectal Cancer Metastatic; Colorectal Cancer
Keywords: IVLP; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVLP in single lung (Experimental)
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin infusion in single lung via IVLP technique

SUMMARY:
This study is investigating a new technique for delivering chemotherapy directly into the lungs at the time of surgery. Delivering chemotherapy directly to the lungs could potentially kill any microscopic cancer cells that are present in the lungs at the time of surgery, while sparing other major organs in the body from the side effects of chemotherapy. This technique is called In Vivo Lung Perfusion (IVLP). At the University Health Network, this IVLP technique has been used recently in a Phase I study in patients with sarcoma, and we are now expanding on that experience to include patients with colorectal metastases. The purpose of this study is to test the safety of the IVLP technique and find the dose that seems right in humans. Participants are given oxaliplatin into one lung via IVLP and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then more participants are asked to join the study and are given a higher dose of oxaliplatin. Participants joining the study later on will get higher doses of oxaliplatin than participants who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given. The other lung will not be infused with anything, so that we can limit unforeseen toxicity to a single lung and see if one lung does better than the other.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Colorectal Carcinoma
2. Presence of bilateral pulmonary metastases
3. 3 or more lung lesions in total
4. Age 70 years or less
5. ECOG 0-2
6. Absence of extra-pulmonary disease, except liver metastases suitable to curative treatment.

Exclusion Criteria:

1. Patient has previously received more than 1000 mg of oxaliplatin
2. Left Ventricular Ejection Fraction <50%
3. History of significant pulmonary disease or pneumonitis
4. Pregnant or lactating females
5. Age 71 or older, or less than 18 years
6. Inability to understand the informed consent process
7. Hypersenstivity to oxaliplatin
8. Patients with Heparin-induced thrombocytopenia (HIT)
9. Patients who cannot receive cefazolin or methylprednisolone due to allergy or another reason can be included but will not receive the drug they cannot tolerate
10. Current participation in another therapeutic clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
safety as measured by acute lung injury findings | 72 hours
  Chest x- ray findings of pulmonary edema in the perfused lung in the first 72 hours (Grade 0-5).

SECONDARY OUTCOMES:
recurrence patterns | 5 years
Incidence of pneumonia after procedure | 72 hours
Incidence of ICU admission | 72 hours
Incidence of mechanical ventilation | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo K Cypel, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No